CLINICAL TRIAL: NCT02043756
Title: Phase I and Pharmacokinetic Study of Mitoxantrone Hydrochloride Liposome Injection in Patients With Solid Tumor
Brief Title: Phase I and Pharmacokinetic Study of Mitoxantrone Hydrochloride Liposome Injection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: cspcmitlip
Record Dates: First submitted 2014-01-16; First posted 2014-01-23 (Estimated); Last update posted 2014-01-23 (Estimated); Status verified 2014-01

CONDITIONS: Neoplasms
Keywords: Mitoxantrone Hydrochloride Liposome Injection
MeSH Terms: conditions — Neoplasms | interventions — Mitoxantrone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mitoxantrone Hydrochloride Liposome (Experimental): Dose escalation will begin at 6mg/m2 to 16mg/m2,4 weeks apart
  Interventions: Drug: Mitoxantrone Hydrochloride Liposome
- Mitoxantrone ,injection (Active Comparator): When the dose of experiment drup up 10mg/m2,10mg/m2 of Mitoxantrone as active comparator
  Interventions: Drug: Mitoxantrone

INTERVENTIONS:
Drug: Mitoxantrone Hydrochloride Liposome — 6-16mg/m2, IV ,one time of each 28 day cycle,3 cycles
  Other Names: 2010L04017
  Arms: Mitoxantrone Hydrochloride Liposome
Drug: Mitoxantrone — 10mg/m2, IV ,on day 1 of each 28 day,3 cycles
  Other Names: Novantrone
  Arms: Mitoxantrone ,injection

SUMMARY:
The purpose of the study is to examine the toxicity profile, maximum tolerated dose (MTD), and pharmacokinetics of Mitoxantrone Hydrochloride Liposome Injection.

DETAILED DESCRIPTION:
The trial of the dose escalation method is from the minimum dose until the maximum tolerated dose and every 3 patient is a dose group.

ELIGIBILITY:
Inclusion criteria:

* Patients must compliance with the requirements and restrictions listed in the consent form
* Patients with Pathology and / or cytologically proven malignant solid tumor
* Patients must be 18-70 years old ,both male and female
* Failure of standard chemotherapy
* Patients have no better choice and may be benefit from the use of anthracyclines
* Patients must have Eastern Cooperative Oncology Group (ECOG)Performance Status of 0-2
* Objective tumor from the last chemotherapy, biological therapy or other experimental interval treatment least 4 weeks
* Expected survival time ≥ 3 months
* Patients agreed to take effective contraceptive measures during the trial
* Blood routine, liver and kidney function, cardiac function examination in accordance with the following requirements.

Exclusion criteria:

* Pregnancy and breast-feeding women
* Multiple sclerosis
* Patients that have histories of ischemic heart disease and heart congestive,arrhythmia that need to be a treatment and significant valvular disease
* Patients with heart disease induced by anthracycline
* Patients requiring other antineoplastic treatment
* Patients with temperature above 38 degrees or active infection that may effects in clinical tests
* Patients are allergic to anthracycline and liposomal drugs
* Patients are allergic to eggs,egg products,soybean and soybean products
* Patients with uncontrolled primary or metastatic brain tumors

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-08; Primary Completion 2013-06 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
To determination the maximal tolerance dose and dose-limiting toxicity of Mitoxantrone Hydrochloride Liposome | 3 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yuankai Shi, Ph.D, Principal Investigator — Cancer Hospital ,Chinese Academy of Mddical Sciences 010-87788701; Jianliang Yang, Ph.D, Study Director — Cancer Hospital ,Chinese Academy of Mddical Sciences 010-87788121; Xiaohong Han, Ph.D, Study Director — Cancer Hospital ,Chinese Academy of Mddical Sciences 010-87788701

REFERENCES:
- [Derived] Yang J, Shi Y, Li C, Gui L, Zhao X, Liu P, Han X, Song Y, Li N, Du P, Zhang S. Phase I clinical trial of pegylated liposomal mitoxantrone plm60-s: pharmacokinetics, toxicity and preliminary efficacy. Cancer Chemother Pharmacol. 2014 Sep;74(3):637-46. doi: 10.1007/s00280-014-2523-8. Epub 2014 Jul 18. PMID 25034977